CLINICAL TRIAL: NCT04913545
Title: The Senstivity and Specificity of Using Salivary Extracellular Vesicles as Non -Invasive Source of miRNAs (412,512) in Detection of Malignant Transformation of Potientially Malignant Oral Lesions.
Brief Title: The Senstivity and Specificity of Using Salivary miRNAs in Detection of Malignant Transformation of Oral Lesions.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Neveen Nabil Ghareeb, assistant lecturer in MSA university, Cairo University
Other Study IDs: 19 September,2018 ,Version 2
Record Dates: First submitted 2021-05-29; First posted 2021-06-04 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Oral Premalignant Lesions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- normal group: participants with out any systemic medical problemes or oral lesions. we will only take saliva sample.
  Interventions: Diagnostic Test: using salivary miRNA (412,512)
- potientially malignant group: participants with suspicious oral lesions without any medical diseases. we will take saliva sample and take a biopsy sample .
  Interventions: Diagnostic Test: using salivary miRNA (412,512)
- malignant group: participants with already diagnosed oral malignant lesions without receiving any treatment yett
  Interventions: Diagnostic Test: using salivary miRNA (412,512)

INTERVENTIONS:
Diagnostic Test: using salivary miRNA (412,512) — quantitative real time polymerase chain reaction to detect the salivary miRNAs 412,512) to indicate the malignant transformation in potientially malignant oral lesions.
  Other Names: biopsy sample for potientially maliganat and malignant group

SUMMARY:
Due to cancer is a leading cause of death world wide , we will coduct the study to evaluate the diagnostic accuracy of using salivary miRNAs (412,512) from the salivary extracellular vesicles (index test) in detection of the malignant transformation of the premalignant lesions using the qualitative real time polymerase chain reaction (qRT-PCR) analysis in comparison to taking biopsy .

DETAILED DESCRIPTION:
our study is a case control study,we will coduct our study to evaluate specificity and sensitivity of using salivary extracellular vesicles miRNAs (412,512) in detection of malignant transformation in potientially malignant oral lesions by using qRT-PCR analysis ,participants will be selected and arranged in 3 groups the control group, potentially malignant group and malignant group ,the salivary samples from the participants will be collected and then microRNA extraction steps will be done through the laboratory steps ,that include extracellular vesicles isolation, PCR Analysis for miRNA-412 and miRNA-512 expression ,also the histopathologic diagnosis and examination of all specimens were confirmed by pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Clinically evident lesions as morphologically altered tissue noted at conventional visual tactile examination
* Clinically evident suspicious lesions which are morphologically altered tissue noted at comprehensive visual ductile examination ( CVTE) with a definitive diagnosis of a potentially malignant disorders (PMD) or even a malignant disorder to be a distinct possibly.
* Healthy subjects presenting no clinically detectable oral lesions matched for age, gender, and risk factors will recruited as controls.

Exclusion Criteria:

.<18 years of age.

* pregnant or breast feeding. .psychiatrically or mentally unstable.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group of normal control subjects: 18 Healthy subjects presenting no clinically detectable oral lesions matched for age, gender, and risk factors .Group of subjects with potentially malignant lesions: 18 patient with innocuous lesions.
  * Group of subjects with malignant lesions:18 patient with suspicious lesions
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
the sensitivity and specificity of salivary miRNAs (412,512) to detect the malignant transformation of oral potentially malignant lesions | 2 years
  measuring the sensitivity and specificity of using the salivary miRNAs(412,512)to detect the malignant transformation in potentially malignant lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ghareeb, Principal Investigator — Assistant lecturer
Locations (1):
- Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided